CLINICAL TRIAL: NCT01130922
Title: Pharmacokinetic Evaluation of Moxifloxacin Administered Intravenously and Orally in Healthy Volunteers Who Have Had a Gastric Bypass.
Acronym: DRUG10_MOXI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Jan Van Bocxlaer, PhD, University Ghent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010/099
Record Dates: First submitted 2010-04-22; First posted 2010-05-26 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Gastric Bypass; Body Weight
Keywords: Roux-and-Y gastric bypass surgery; stable body weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin IV (Experimental)
  Interventions: Drug: moxifloxacin per IV
- Moxifloxacin oral (Active Comparator)
  Interventions: Drug: moxifloxacin per os

INTERVENTIONS:
Drug: moxifloxacin per IV — intravenous administration of 400 mg moxifloxacin (as a 1h-infusion)
  Arms: Moxifloxacin IV
Drug: moxifloxacin per os — oral administration of 400 mg moxifloxacin in a single dose
  Arms: Moxifloxacin oral

SUMMARY:
Roux-and-Y gastric bypass is one of the most common forms of bariatric surgery; due to a reduction in size of the stomach and intestine, the available surface area for the absorption of oral drugs is strongly decreased. This may lead to a reduced bioavailability resulting in a reduced efficacy of the drug. However, in literature there is no information available about the impact of bariatric surgery on the pharmacokinetics of moxifloxacin. This protocol evaluates the moxifloxacin plasma levels, the variability between subjects and the absolute bioavailability, after oral administration of 400 mg moxifloxacin in healthy volunteers who have had a gastric bypass at least 6 months ago and who now have a stable body weight.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who have had a gastric bypass at least 6 months ago and whose body weight has not changed more than 5% during the last 3 months
* Age between 18 and 60 years old
* Able to give informed consent

Exclusion Criteria:

* Other forms of bariatric surgery (Scopinaro and Mason/Sleeve) before gastric bypass surgery
* Hypersensitivity to moxifloxacin, other quinolones or to any of the excipients
* Pregnancy and lactation
* Creatinine clearance < 80 ml/min
* Transaminases > 2x the upper limit of normal (AST/ALT)
* Impaired liver function (Child Pugh C)
* Fasting glycaemia > 125mg/dl
* Epilepsy
* Patients with a history of tendon disease/disorder (especially Achilles tendon rupture) related to quinolone treatment
* Patients with the following heart disorders:

  * Electrolyte disturbance, particularly an uncorrected hypokalaemia
  * Clinically relevant bradycardia
  * Clinically relevant heart failure with reduced left-ventricular ejection fraction
  * Previous history of symptomatic arrhythmias
* Congenital or documented acquired QT prolongation or concurrently use of drugs that prolong the QT interval:

  * anti-arrhythmics (Classes IA and III)
  * neuroleptics
  * tricyclic antidepressants
  * antimicrobials (e.g. sparfloxacin, intravenous erythromycin, pentamidine, antimalarials particularly halofantrine)
  * some antihistamines (e.g. terfenadine, astemizole, mizolastine)
  * cisapride, intravenous vincamine, bepridil and diphemanil
* No normal thyroid function
* All clinically significant disorders that can interfere with the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of 400 mg moxifloxacin per IV compared to 400 mg moxifloxacin per os in patients who had a gastric bypass | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van Bocxlaer, PhD, Principal Investigator — University Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] De Smet J, Colin P, De Paepe P, Ruige J, Batens H, Van Nieuwenhove Y, Vogelaers D, Blot S, Van Bocxlaer J, Van Bortel LM, Boussery K. Oral bioavailability of moxifloxacin after Roux-en-Y gastric bypass surgery. J Antimicrob Chemother. 2012 Jan;67(1):226-9. doi: 10.1093/jac/dkr436. Epub 2011 Oct 10. PMID 21987240